CLINICAL TRIAL: NCT03850639
Title: An Internet-delivered Cognitive-behavioral Intervention Provided Soon After Trauma: a Two-step Feasibility Trial
Brief Title: An Internet-delivered Cognitive-behavioral Intervention Provided Soon After Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2018/2365-31
Record Dates: First submitted 2019-02-15; First posted 2019-02-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The experimental group will go through active internet-based treatment which is delivered on a safe internet platform. Treatment is divided into four modules, each containing homework assignments. Participants in experimental group will be assigned a therapist that they can contact through a message system in the platform and expect answer within 48 hours.
Masking Description: Waitlist control, i.e. no active active intervention during waiting list period. Will be offered treatment after 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based exposure therapy (Experimental): The experimental group will go through active internet-based treatment which is delivered on a safe internet platform. Treatment is divided into four modules, each containing homework assignments. Participants in experimental group will be assigned a therapist that they can contact through a message system in the platform and expect answer within 48 hours.
  Interventions: Behavioral: Internet-based exposure therapy
- Wait list control (No Intervention): Waitlist control, i.e. no active active intervention during waiting list period. Will be offered treatment after 4 weeks.

INTERVENTIONS:
Behavioral: Internet-based exposure therapy — The treatment is a three week long cognitive behavior therapy. It is based mainly on the principles of exposure; i.e. the participant is instructed to approach the memory of the traumatic event and situations they since the traumatic events are associated with fear and anxiety. Other interventions include psychoeducation, and breathing retraining to facilitate exposure.
  Arms: Internet-based exposure therapy

SUMMARY:
The primary objective with this study is to investigate the feasibility of an internet-delivered cognitive-behavioral (CBT) intervention provided soon after trauma (within 2 months). The secondary objective is to investigate the effects of the internet-delivered CBT intervention on intrusive memories compared to no treatment.

DETAILED DESCRIPTION:
Objective The primary objective with this study is to investigate the feasibility of an internet-delivered psychological intervention provided soon after trauma (within 2 months). The secondary objective is to investigate the effects of the internet-delivered CBT intervention on intrusive memories compared to no treatment.

Trial design We will first pre-pilot test the intervention- and assessment procedures in five participants (no randomization) which will be followed by a randomized controlled trial with waitlist control. The wait list control group will also receive treatment after the first group has finished.

SAMPLE SIZE 5 plus 30 participants.

ENDPOINTS Self-report assessment of daily intrusions at baseline and post-treatment

SECONDARY ENDPOINTS The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) at baseline (and post-treatment Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) at baseline and post-treatment.

Euroqol, EQ-5D at baseline and post-treatment.

Recruitment Self-referral. Advertising will be made through national newspapers, social media, patient organisations' and ads directed to health care units, such as emergency departments, in Sweden.

Safety parameters Participants will have the opportunity to report any adverse events during treatment at posttreatment and follow-up measurements.

Data collection: Data will be collected electronically via the treatment platform and a safe app.

Main statistical analysis:

Between-group estimates on outcome are done using a mixed-effects regression model with a Poisson distribution. All analyses will be done according to intention to treat and post hoc per protocol analyses will also be conducted. The primary criterion is the estimated regression slope of daily intrusive memories between day 0-7 and day 28-35.

ELIGIBILITY:
Inclusion Criteria:

* Experienced psychological trauma according to criterium A for PTSD in the DSM-5 (exposed to death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence) the past two months.
* Ongoing intrusive memories from this traumatic event
* ≥ 18 years
* Situated in Sweden
* Informed consent

Exclusion Criteria:

* Other serious comorbidity as primary concern (ongoing substance dependence, untreated bipolar disorder, psychotic symptoms, severe depression, borderline personality disorder, high suicidal risk according to the MINI)
* Not fluent speaking in Swedish
* Receiving CBT for trauma
* Ongoing trauma-related threat (e.g. living with a violent spouse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-12-02 (Estimated); Study Completion 2021-06-05 (Estimated)

PRIMARY OUTCOMES:
Number of intrusion of the traumatic memory | Baseline (day 0-7), post-treatment (day 28-35) and follow-up 6 months
  Change in self-report assessment of daily intrusions at baseline (day 0-7) and post-treatment (day 28-35). The participants are each day asked to report number of intrusive memories during morning, afternoon, evening and night through a smart phone app. If the participants don't have access to a smart phone, pen and stencil will be used.

SECONDARY OUTCOMES:
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline (day 0-7), post-treatment (day 28-35) and follow-up 6 months
  Change in symptoms of post traumatic stress from baseline to post treatment and follow up (6 months). The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. All items are scored on a 0-4 scale. Higher score indicate worse severity.
Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) | Baseline (day 0-7), post-treatment (day 28-35) and follow-up 6 months
  Change in depressive symptoms from baseline to post treatment and follow up (6 months). The Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) is a 9 item self-report measure that assesses the presence and severity of depressive symptoms. All items are scored on a 0-6 scale. Higher score indicate worse severity.
Euroqol, EQ-5D | Baseline (day 0-7), post-treatment (day 28-35) and follow-up 6 months
  Change in overall health from baseline to post treatment and follow up (6 months). EQ-5D is a standardised self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Andersson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bragesjo M, Arnberg FK, Andersson E. Mediators of change in a condensed online exposure-based intervention provided soon after trauma: insights from a randomised controlled trial. Eur J Psychotraumatol. 2024;15(1):2430807. doi: 10.1080/20008066.2024.2430807. Epub 2024 Dec 2. PMID 39621100